CLINICAL TRIAL: NCT07157865
Title: A Comparison of Prism Adaptation Training (PAT) Paired With Transcutaneous Electrical Stimulation (TENS) vs PAT Alone on Outcomes in Post-Stroke Patients Experiencing Unilateral Spatial Neglect (USN)
Brief Title: Comparing Prism Adaptation Training With and Without TENS to Minimize Unilateral Spatial Neglect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHN-2025-113
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Unilateral Spatial Neglect; Stroke
MeSH Terms: conditions — Stroke | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PAT + TENS treatment (Experimental): Subjects in this group will receive both prism adaptation training (PAT) and transcutaneous electrical nerve stimulation (TENS) during therapy sessions. Subjects will wear 20 diopter prism lenses that shift the visual field (for left neglect field is shifted to right, for right neglect field is shifted to the left) while reaching with either UE toward a target. The visual system and the motor system adapt over several reaches to align both the visual system and the motor system, and the target is reached. The client will wear the prism goggles during the functional reaching task while also using a TENS unit on their upper extremity on the neglected side of space to provide increased sensory awareness. TENS will be delivered using FDA-approved commercially available portable units.
  Interventions: Device: Prism adaptation training combined with TENS
- PAT only (Active Comparator): Subjects will receive only prism adaptation training (PAT) during their therapy sessions. Subjects will wear 20 diopter prism lenses that shift the visual field (for left neglect field is shifted to right, for right neglect field is shifted to the left) while reaching with either UE toward a target. The visual system and the motor system adapt over several reaches to align both the visual system and the motor system, and the target is reached. The client will wear the prism goggles during the functional reaching task.
  Interventions: Other: PAT only

INTERVENTIONS:
Device: Prism adaptation training combined with TENS — Subjects in the experimental group will receive both prism adaptation training and TENS to identify affects on USN. To date there are no published studies combining these treatments to minimize USN.
  Arms: PAT + TENS treatment
Other: PAT only — Subjects will receive prism adaptation training (PAT) only wearing prism goggles during a functional reaching task during occupational therapy.
  Arms: PAT only

SUMMARY:
This study aims to find out if doing two treatments together-Prism Adaptation Therapy (PAT) and Transcutaneous Electrical Nerve Stimulation (TENS)-will help people who have had a stroke pay better attention to one side of their body, better than just doing PAT by itself.

In addition to understanding how the intervention improves function the investigators would like to see if things like how old someone is, how long ago their stroke happened, where their brain was damaged, or how bad the neglect is, affect how well the treatment works.

To measure if the interventions make a difference the following outcome measures will be used.

Catherine Bergego Scale (CBS):

This is a test to see how severe someone's neglect is. Trained therapists use 10 simple tasks to check if a person is ignoring the left or right side.

Wolf Motor Function Test (WMFT):

This test checks how well a stroke survivor can move their arm. It helps the therapists see if the treatments improve movement and reaction time

People can join the study if they had a stroke, score at least "1" on the Catherine Bergego Scale, and they can understand and agree to take part in the study.

People cannot join the study if they have had more than two strokes, have or had seizures, or have a serious mental illness like schizophrenia, or have cancer in the arm that was affected by the stroke, they have a pacemaker or defibrillator in their body, and if they can't feel their arm on the side affected by the stroke

Once the study is done, the main results will be shared with the therapists who work at the NeuroRehab and Balance Center, like the physical, speech, and occupational therapists.

DETAILED DESCRIPTION:
Unilateral spatial neglect (USN) is a common and disabling consequence of stroke, particularly following right-hemisphere lesions, affecting up to 50-70% of survivors. USN impairs a patient's ability to attend to or interact with stimuli on the side opposite the brain lesion, leading to significant challenges in daily functioning and rehabilitation engagement. The presence of USN is associated with poorer functional outcomes, increased dependence, and prolonged recovery after a stroke. Prism Adaptation Training (PAT) is a non-invasive intervention that has emerged as a promising approach for USN rehabilitation. PAT involves repeated visuomotor activities while wearing prism glasses that shift the visual field, promoting adaptation and recalibration of spatial attention. Multiple studies and systematic reviews have demonstrated that PAT can improve neglect symptoms, enhance motor control of the affected limb, and improve activities of daily living (ADL), with effects persisting for weeks to months post-intervention. However, the optimal dosing, duration, and potential for augmenting the effects of PAT remain areas of ongoing investigation. Transcutaneous Electrical Nerve Stimulation (TENS) is another non-invasive modality widely used in post-stroke rehabilitation. TENS delivers mild electrical currents through the skin to stimulate nerves and has shown efficacy in improving motor function, reducing spasticity, and enhancing functional recovery in stroke survivors. It has been shown to enhance upper limb function in individuals who have experienced a stroke. While TENS is primarily used for motor and sensory rehabilitation, its potential to modulate cortical excitability and facilitate neuroplasticity suggests it may also influence cognitive domains, including attention and spatial processing. There is evidence suggesting that TENS can have an impact on neglect. Despite the individual benefits of PAT and TENS in post-stroke rehabilitation, limited research has explored their combined effects on USN. The rationale for pairing PAT with TENS is based on the hypothesis that TENS-induced sensory stimulation may help enhance awareness of neglected space when applied to the upper extremity of individuals experiencing neglect, thereby potentially amplifying the adaptive effects of PAT on spatial neglect. However, the synergistic potential of TENS to enhance cognitive-perceptual rehabilitation strategies like PAT in the context of USN has not been systematically investigated. Given the persistent functional burden of USN and the need for more effective and accessible rehabilitation protocols, a pilot study comparing PAT paired with TENS versus PAT alone could provide critical preliminary evidence. Such research may identify whether adjunctive TENS can accelerate or enhance recovery from neglect, inform optimal intervention strategies, and ultimately improve independence and quality of life for stroke survivors experiencing USN.

The research question:

Is the combination of Prism Adaptation Therapy (PAT) and Transcutaneous Electrical Nerve Stimulation (TENS) more effective than PAT alone in reducing unilateral spatial neglect (USN) in individuals' post-stroke?

Hypothesis: The combination of Prism Adaptation Therapy (PAT) and Transcutaneous Electrical Nerve Stimulation (TENS) will be more effective than PAT alone in reducing unilateral spatial neglect (USN) in individuals post-stroke.

Primary study aim:

To evaluate whether the combination of Prism Adaptation Therapy (PAT) and Transcutaneous Electrical Nerve Stimulation (TENS) is more effective than PAT alone in reducing unilateral spatial neglect (USN) in individuals post-stroke.

Secondary study aims: To investigate whether patient characteristics (e.g. time since stroke, lesion location, severity of neglect, gender, age) influence the effectiveness of the combined intervention. To investigate the effects of the PAT alone and the combined PAT and TENS intervention on functional outcomes related to USN. To investigate the impact of PAT alone and the combined PAT and TENS intervention on the motor control of the neglected limb.

The main study outcome measures include:

The Catherine Bergego Scale (CBS) is the selected outcome measure for assessing the severity of Unilateral Spatial Neglect (USN) and for evaluating changes in function and neglect following interventions. The CBS includes 10 subtests designed to identify both the presence and severity of USN. All occupational therapists at the NeuroRehab and Balance Center (NRBC) have been trained in the proper administration and scoring of the CBS to ensure accurate results. It is standard protocol at NRBC clinic that all patients diagnosed with stroke are evaluated for potential USN using the CBS, which is routinely administered in these cases. In 2014, the Kessler Foundation published guidelines on how to administer the CBS.

The Wolf Motor Function Test (WMFT) is a standardized assessment tool widely used to measure upper extremity motor abilities in individuals recovering from a stroke. This test serves as an outcome measure for motor control, helping to assess improvements in movement quality and reaction time following interventions. All occupational therapists at the NeuroRehab and Balance Center (NRBC) have received training in the administration and scoring of the WMFT, and it is standard protocol at NRBC that all patients diagnosed with stroke are evaluated using the WMFT.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of stroke
* Score 1 or above on the Catherine Bergego Scale
* Cognitively able to consent

Exclusion Criteria:

* Seizure disorder
* Diagnosed with more than two strokes
* Diagnosis of schizophrenia or schizoaffective disorder
* Cancer diagnosis of upper extremity
* Individuals with pacemakers and debrillators
* Absent sensation of upper extremity affected by stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in unilateral spatial neglect functional deficits | From enrollment to discharge from therapy services which is typically 8-12 weeks
  The Catherine Bergego Scale (CBS) is the selected outcome measure for assessing the severity of Unilateral Spatial Neglect (USN) and for evaluating changes in function and neglect following interventions. The CBS includes 10 subtests designed to identify both the presence and severity of USN. Maximum score on the CBS is 30 which indicates severe neglect, minumum score is 0 which indicates no neglect.
Change in motor control deficits | From time of enrollment to discharge from therapy services typically 8-12 weeks
  The Wolf Motor Function Test (WMFT) is a standardized assessment tool widely used to measure upper extremity motor abilities in individuals recovering from a stroke. This test serves as an outcome measure for motor control, assessing motor ability via a performance time and a Functional Ability Scale (FAS) of 15 subtests. During the timed tests subjects are allowed a maximum of 120 seconds per task. If a person cannot complete the task within 120 seconds the time is recorded as 120+. The official WFMT time score is the median time of 15 timed tasks. The FAS is calculated using a 6-point ordinal scale from 0-5. A higher score indicates better movement (0 = does not attempt to use the affected limb to 5=movement appears normal). The FAS score is calculated by averaging scores across all subtests.

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle M Janning, OTD, MS, OTR/L, Principal Investigator — Kettering Health/Northern Kentucky University
Locations (1):
- Kettering Health NeuroRehab and Balance Center, Centerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share age, sex, gender, and time since stroke of research subjects. Statistical analysis results summary including primary outcomes.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from December 15, 2027 to May 15, 2028
Access Criteria: Data will be shared by the principle investigator by request for data analysis to address research questions.

REFERENCES:
- [Background] Song C, Wu W, Feng N, Li Z, Lei B. Rehabilitative effects of Transcutaneous Electric Nerve Stimulation on limb function in stroke patients: a systematic review and meta-analysis. Disabil Rehabil. 2025 Sep;47(18):4645-4652. doi: 10.1080/09638288.2025.2453640. Epub 2025 Feb 11. PMID 39930993
- [Background] Jacquin-Courtois S, O'Shea J, Luaute J, Pisella L, Revol P, Mizuno K, Rode G, Rossetti Y. Rehabilitation of spatial neglect by prism adaptation: a peculiar expansion of sensorimotor after-effects to spatial cognition. Neurosci Biobehav Rev. 2013 May;37(4):594-609. doi: 10.1016/j.neubiorev.2013.02.007. Epub 2013 Feb 18. PMID 23428624
- [Background] Fortis P, Ronchi R, Velardo V, Calzolari E, Banco E, Algeri L, Spada MS, Vallar G. A home-based prism adaptation training for neglect patients. Cortex. 2020 Jan;122:61-80. doi: 10.1016/j.cortex.2018.09.001. Epub 2018 Sep 18. PMID 30314612
- [Background] Eslami, S., Tahmasbi, F., Mohammadzadeh, S., Sanaie, S., Ghaderi, S., & Mamaghani, A.R.(2024). Application of transcutaneous electrical nerve stimulation (TENS) in stroke rehabilitation: An umbrella review. NeuroRegulation, 11(3), 304-325. doi:10.15540/nr.11.3.304
- [Background] Chen P, Hreha K, Gonzalez-Snyder C, Rich TJ, Gillen RW, Parrott D, Barrett AM. Impacts of Prism Adaptation Treatment on Spatial Neglect and Rehabilitation Outcome: Dosage Matters. Neurorehabil Neural Repair. 2022 Aug;36(8):500-513. doi: 10.1177/15459683221107891. Epub 2022 Jun 8. PMID 35673990
- [Background] Chen P, Diaz-Segarra N, Hreha K, Kaplan E, Barrett AM. Prism Adaptation Treatment Improves Inpatient Rehabilitation Outcome in Individuals With Spatial Neglect: A Retrospective Matched Control Study. Arch Rehabil Res Clin Transl. 2021 May 19;3(3):100130. doi: 10.1016/j.arrct.2021.100130. eCollection 2021 Sep. PMID 34589681
- [Background] Chen, P., et al. (2015). Relationship between visual neglect and rehabilitation outcomes in stroke patients: A meta-analysis. American Journal of Physical Medicine & Rehabilitation, 94(7), 567-578.
- [Background] Champod AS, Frank RC, Taylor K, Eskes GA. The effects of prism adaptation on daily life activities in patients with visuospatial neglect: a systematic review. Neuropsychol Rehabil. 2018 Jun;28(4):491-514. doi: 10.1080/09602011.2016.1182032. Epub 2016 May 16. PMID 27181587